CLINICAL TRIAL: NCT00771186
Title: Intraoperative Laryngeal Electromyography (LEMG) in Children With Vocal Fold Immobility: a Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Christopher Hartnick MD, Massachusetts Eye and Ear Infirmary
Other Study IDs: 07-12-078x
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Vocal Fold Immobility
Keywords: pediatric; Laryngeal EMG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children with vocal fold immobility

SUMMARY:
The goal of this study is to further study the role of LEMG in accurately predicting the recovery of vocal function as well to study the timing of a change of LEMG activity prior to such return of function. We aim to do this by collaborating with several active pediatric otolaryngological practices throughout the country who in turn have agreed to evaluate infants and children with vocal fold immobility who fit a standardized inclusion and exclusion criteria by means of a standardized LEMG protocol over a one year period of time. Our particular goal is to collect and then review information over a one year period of time on all children evaluated for vocal fold immobility by means of LEMG.

DETAILED DESCRIPTION:
Study design:

Primary central hypothesis:

Operative LEMG performed in a serial fashion can predict return of RLN function in children after iatrogenic injury.

Secondary hypothesis:

Operative LEMG performed in a serial fashion will allow some projection as to the timing of RLN recovery

Inclusion criteria:

1. Children age 0-18 with vocal fold immobility documented by laryngeal fiberoptic evaluation
2. Children who have had a recent, identifiable cardiac surgical etiology for RLN injury and subsequent VFI
3. Children whose parents sign informed consent and who themselves sign assent if they are old enough to do so.

Exclusion criteria

1. Children whose families do not give informed consent or who themselves do not give informed assent ( if the children are old enough to understand)
2. Children with congenital VFI where the etiology is not clearly identified

Data to be recorded:

1. Age of patient
2. Gender
3. Age of initial fiberoptic evaluation and of initial diagnosis
4. Diagnosis
5. Serial Laryngeal Recordings
6. Fiberoptic Evaluations

LEMG Recording

While in a light plane of anesthesia, the following recordings will be routinely performed:

1. 10 seconds of both right and left vocal fold LEMG simultaneously recorded with a gain of 50 V
2. 10 seconds of both right and left vocal fold LEMG simultaneously recorded with a gain of 200 V
3. 10 seconds of right vocal fold LEMG recorded with a gain of 50 V
4. 10 seconds of right vocal fold LEMG recorded with a gain of 200 V
5. 10 seconds of left vocal fold LEMG recorded with a gain of 50 V
6. 10 seconds of left vocal fold LEMG recorded with a gain of 200 V

Total recording time: 60 seconds

Timing of LEMG and Awake Fiberoptic Laryngoscopy

Following current standard clinical evaluation we are performing at MEEI, we propose to perform awake fiberoptic laryngoscopy and operative LEMG at the following time points: initially (within 3 weeks of injury if possible), at the 3 month post-injury mark, and at the 9- month post injury mark ( 3 recordings in total; we will perform a final fiberoptic laryngoscopy in the office at the one year time interval). The time points were chosen as each recording necessitates an operative procedure with general anesthesia so we wanted to limit the over number of general anesthetics. We recognize that the risk of limiting the number of operative LEMG recordings is that we lose some data-points to chart recovery of RLN function, but we felt that the risks of multiple general anesthetics were sufficient enough to warrant limiting the number of recordings as much as possible.

Data Collection and Database protection

All Data collected will be entered into a password protected database.

ELIGIBILITY:
Inclusion Criteria:

1. Children age 0-18 with vocal fold immobility documented by laryngeal fiberoptic evaluation
2. Children who have had a recent, identifiable cardiac surgical etiology for RLN injury and subsequent VFI
3. Children whose parents sign informed consent and who themselves sign assent if they are old enough to do so

Exclusion Criteria:

1. Children whose families do not give informed consent or who themselves do not give informed assent ( if the children are old enough to understand)
2. Children with congenital VFI where the etiology is not clearly identified

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with vocal fold immobility
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
return of vocal fold function | one year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Maturo SC, Braun N, Brown DJ, Chong PS, Kerschner JE, Hartnick CJ. Intraoperative laryngeal electromyography in children with vocal fold immobility: results of a multicenter longitudinal study. Arch Otolaryngol Head Neck Surg. 2011 Dec;137(12):1251-7. doi: 10.1001/archoto.2011.184. PMID 22183907